CLINICAL TRIAL: NCT01833078
Title: Ghrelin in Frail Elderly Subcutaneous Repeated Dose Study
Brief Title: Ghrelin Repeated Dose Study
Acronym: GRD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Anne Cappola, Associate Professor of Medicine, Perelman School of Medicine, University of Pennsylvania
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 817283
Record Dates: First submitted 2013-04-11; First posted 2013-04-16 (Estimated); Results first posted 2015-10-08 (Estimated); Last update posted 2015-10-08 (Estimated); Status verified 2015-09

CONDITIONS: Frailty in Aging
MeSH Terms: interventions — Ghrelin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 7 day ghrelin dosing - all participants (Other): All participants will receive an injection of ghrelin (7.5mcg/kg) dose subcutaneously once daily on Days 1, 2 and 7 in the research center and will self-administer the subcutaneous injection before breakfast on Days 2-6 at home.
  Interventions: Drug: ghrelin

INTERVENTIONS:
Drug: ghrelin — ghrelin administration subcutaneously for 7 days

SUMMARY:
Frailty is a geriatric syndrome leading to physical deterioration including muscle wasting (sarcopenia) and unintentional weight loss. There are currently no approved therapies for frailty. Ghrelin is a hormone produced by the stomach that stimulates appetite centers in the brain. The investigators already know that a single dose of Ghrelin improves food intake immediately after the dose in frail older people. In this study, the investigators are trying to find out if repeated daily doses of ghrelin will help frail older people improve food intake for multiple days in a row.

DETAILED DESCRIPTION:
The study design is an open label, repeated dose administration study in which we will examine the safety and efficacy of repeated subcutaneous ghrelin administration in frail individuals. There will be a screening visit plus three additional study visits at the CTRC on Days 1, 2, and 7. Participants will receive an injection of ghrelin subcutaneously once daily on Days 1 and 7 and will self-administer the subcutaneous injection before breakfast on Days 2-6 at home. A food record will be kept from Day -3 to Day 6. We will assess the efficacy of repeated ghrelin doses to sustainably increase caloric intake from pre-treatment baseline without hyperglycemia or raising of cortisol levels.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with three, four or five frailty criteria using the Fried frailty criteria

Exclusion Criteria:

1. Diabetes mellitus or fasting glucose ≥ 126 mg/dL
2. Hospitalization for stroke, myocardial infarction, coronary artery bypass graft surgery, vascular surgery in the past six months.
3. New York Heart Association Class III or IV congestive heart failure
4. Therapy for cancer in the past 12 months, except non-melanoma skin cancer
5. BMI ≥ 30 kg/m2
6. Current use of corticosteroids other than topical, ophthalmic, and inhaled preparations
7. Therapy with megestrol acetate or dronabinol within the last 6 weeks
8. Thyroid stimulating hormone measured as < 0.4 mU/L or greater than 10mU/L
9. Abnormal liver function tests (LFTs > 2x upper limit of normal)
10. Hemoglobin < 11g/dL
11. Insulin-like growth factor-I (IGF-I) above the age-specific reference range
12. History of surgery within the last 30 days
13. Unstable medical or psychological conditions or unstable home or food environment
14. Cognitive deficit as defined by a Folstein Mini Mental State Exam score < 24/30
15. Depression (defined as a score of > 11 on the Geriatric Depression Questionnaire)

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 5 (Actual)
Dates: Start 2013-02; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne Cappola, MD, ScM, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the outpatient medical practice serving the geriatric population at University of Pennsylvania via an electronic alert to physicians. Ten subjects were screened in order to obtain five eligible participants.
Groups:
- Ghrelin: All participants received 7.5 mcg/kg of ghrelin as a once daily subcutaneous dose for seven consecutive days. Days 1, 2 and 7 will be in the research center. Days 3,4,5,and 6 will be self administered at home.
Period: Overall Study
Arm/Group | Ghrelin
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Ghrelin
Number analyzed (Participants) | 5
Age, Continuous [Mean (Full Range); unit: years] | 86 [82 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Safety
Description: 1.Safety: # of participants with treatment emergent adverse events
Time Frame: pre-treatment baseline through 30 days following the last administration of study treatment day 7
Measure: Number; unit: participants
Arm/Group | Ghrelin
Number analyzed (Participants) | 5
participants | 4

2. Secondary Outcome: Sustainability of Increased Caloric Intake
Description: Sustained food intake of standardized meal from Days 1 compared to Day 7.
Time Frame: pre-treatment baseline (day 1) through day 7
Measure: Median (Full Range); unit: calories
Arm/Group | Ghrelin
Number analyzed (Participants) | 5
calories
  Baseline (day 1) | 691 [587 to 1224]
  Day 7 | 839 [548 to 1023]

ADVERSE EVENTS:
Time Frame: Study enrollment through one month following the final visit.
Arm/Group | Ghrelin
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 4/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ghrelin (N=5)
tired (General disorders) | 2
mild diarrhea (Gastrointestinal disorders) | 1
mild and transient abdominal discomfort, rumbling and flatulance (Gastrointestinal disorders) | 1
mild and transient headache (General disorders) | 1
transient feeling of pronounced heartbeat (General disorders) | 1
Mild fatigue (General disorders) | 2
feeling of laziness (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No